CLINICAL TRIAL: NCT04510662
Title: Effectiveness and Safety of Telmisartan in Acute Respiratory Failure Due to COVID-19
Brief Title: Telmisartan in Respiratory Failure Due to COVID-19
Acronym: STAR-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abraham Edgar Gracia-Ramos (Other Government)
Collaborators: National Polytechnic Institute, Mexico (Other)
Responsible Party: Sponsor-Investigator, Abraham Edgar Gracia-Ramos, Physician of the Department of Internal Medicine, Hospital Regional de Alta Especialidad de Zumpango
Organization: Hospital Regional de Alta Especialidad de Zumpango (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI/HRAEZ2020/05
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: COVID-19; Respiratory Insufficiency; Telmisartan; Respiratory Distress Syndrome, Adult
Keywords: COVID-19; telmisartan; respiratory failure; respiratory distress syndrome, adult
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Respiratory Distress Syndrome | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telmisartan (Experimental): Patients in this group will receive telmisartan 40 mg daily plus standard care.
  Interventions: Drug: Telmisartan
- Control (No Intervention): Patients in this group will receive standard care.

INTERVENTIONS:
Drug: Telmisartan — Patients in this group will receive telmisartan 40 mg daily plus standard care.
  Arms: Telmisartan

SUMMARY:
Rationale: The renin-angiotensin-aldosterone system (RAAS) dysregulation may play a central role in the pathophysiology of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection associated acute lung injury (ALI) / acute respiratory distress syndrome (ARDS). In the RAAS, Angiotensin I (Ang I) is converted to angiotensin II (Ang II) by angiotensin converting enzyme (ACE). Ang II mediates vasoconstrictive, pro-inflammatory and pro-oxidative effects through agonism at Ang II type 1 receptor (AT1R). ACE2 converts Ang II to angiotensin 1-7 (Ang1-7), which finally binds to Mas receptor (MasR) and mediates many beneficial actions, including vasodilation and anti-inflammatory, anti-oxidant and antiapoptotic effects. ACE2, a homologue of ACE, is an integral cell membrane protein with a catalytic domain on the extracellular surface exposed to vasoactive peptides. SARS-CoV-2 penetrates the cell through ACE2, and the increase of this receptor (due to the use of ACE inhibitors or angiotensin receptor blockers [ARBs]) may facilitate SARS-CoV-2 infection, which might increase the risk of developing severe and fatal SARS-CoV-2 infection. However, through upregulation of ACE2, ACE inhibitors/ARBs can exert anti-inflammatory and antioxidative effects, which may be beneficial in preventing ALI and ARDS.

Objective: To evaluate the effectiveness and safety of telmisartan in respiratory failure due to COVID-19.

Study design: This is an open label, phase 2 clinical trial. Study population: Adult hospitalized SARS-CoV-2-infected patients (n=60). Intervention: The active-treatment arm will receive telmisartan 40 mg daily and the control arm will receive standard care. Treatment duration will be 14 days or up to hospital discharge <14 days or occurrence of the primary endpoint if <14 days.

Main study endpoint: The primary study endpoint is the occurrence within 14 days of randomization of either: 1) Mechanical ventilation or 2) Death.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age.
* Admitted to the Hospital Regional de Alta Especialidad de Zumpango.
* Confirmed SARS-CoV-2 infection with either: positive laboratory test for SARS-CoV-2; or positive CT thorax diagnostic for SARS-CoV-2 infection according to the prevailing criteria.
* Hypoxic respiratory failure: SpO2 ≤94% on room OR tachypnea (respiratory rate ≥22 breaths/min).

Randomization:

* Within 24 hours of confirmed in-hospital SARS-CoV-2 infection diagnosis OR
* within 24 hours of hospital admission in case of pre-hospital confirmed SARS-CoV-2 infection.
* In case there is a lack of laboratory tests for SARS-CoV-2 in a potentially eligible patient, a positive laboratory test for SARS-CoV-2 will be no longer required. In that case, the potentially eligible patient needs to meet the prevailing criteria for the diagnosis of SARS-CoV-2 infection, such as typical abnormalities on pulmonary CT in the setting of high clinical suspicion of SARS-CoV-2 infection.

Exclusion Criteria:

* Admitted to ICU prior to randomization.
* Currently taking an an angiotensin converting enzyme inhibitor (ACEi) or Angiotensin receptor blocker (ARB).
* Use of other investigational drugs at the time of enrollment
* Prior reaction or intolerance to an ARB; or severe intolerance to an ACEi, defined as angio-oedema requiring medical intervention.
* Systolic blood pressure < 105 mmHg or diastolic blood pressure <65mmHg.
* Potassium greater than 5.5 mEq/L within 4 weeks of study enrollment.
* Estimated Glomerular Filtration Rate (eGFR) of < 30ml/min/1.73 m2 within 4 weeks of study initiation.
* A known history of renal artery stenosis.
* AST and/or ALT > 3 times the upper limit of normal within 4 weeks of study enrollment.
* Severe liver dysfunction (Child-Pugh score C), biliary cirrhosis or cholestasis.
* Severe volume depletion or severe acute kidney injury.
* Inability to obtain informed consent.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Death | Within 30 days
  Death is defined as all-cause mortality
Mechanical ventilation | Within 14 days
  Occurrence of mechanical ventilation

SECONDARY OUTCOMES:
Occurrence of acute kidney injury | Within 14 days
  Defined as a 50% decline in estimated glomerular filtration rate relative to baseline, or decrease of >30 ml/min/1.73m2 and to a value below 60 ml/min/1.73m2
Incidence of hypotension | Within 14 days
  Incidence of episodes of blood pressure less than 90 mm Hg systolic or 60 mm Hg diastolic
Incidence of hypotension requiring vasopressors | Within 14 days
  Outcome reported as the number of participants in each arm requiring the use of vasopressors for hypotension
Incidence of Sepsis | Within 14 days
  Outcome reported as the number of participants in each arm who experience sepsis, defined as the presence of at least 2 of the following clinical criteria together (qSOFA score): respiratory rate of 22/min or greater, altered mentation, or systolic blood pressure of 100 mm Hg or less
Hospital length of stay | Within 14 days
  Hospital length of stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Edgar Gracia-Ramos, MD MSc, Principal Investigator — Hospital Regional de Alta Especialidad de Zumpango
Locations (1):
- Hospital Regional de Alta Especialidad de Zumpango, Zumpango, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers to avoid misuse of patient information.

REFERENCES:
- [Background] Rothlin RP, Vetulli HM, Duarte M, Pelorosso FG. Telmisartan as tentative angiotensin receptor blocker therapeutic for COVID-19. Drug Dev Res. 2020 Nov;81(7):768-770. doi: 10.1002/ddr.21679. Epub 2020 May 1. PMID 32356926
- [Background] Sanchis-Gomar F, Lavie CJ, Perez-Quilis C, Henry BM, Lippi G. Angiotensin-Converting Enzyme 2 and Antihypertensives (Angiotensin Receptor Blockers and Angiotensin-Converting Enzyme Inhibitors) in Coronavirus Disease 2019. Mayo Clin Proc. 2020 Jun;95(6):1222-1230. doi: 10.1016/j.mayocp.2020.03.026. Epub 2020 Apr 4. PMID 32376099
- [Background] Patel AB, Verma A. COVID-19 and Angiotensin-Converting Enzyme Inhibitors and Angiotensin Receptor Blockers: What Is the Evidence? JAMA. 2020 May 12;323(18):1769-1770. doi: 10.1001/jama.2020.4812. No abstract available. PMID 32208485
- [Background] Bavishi C, Maddox TM, Messerli FH. Coronavirus Disease 2019 (COVID-19) Infection and Renin Angiotensin System Blockers. JAMA Cardiol. 2020 Jul 1;5(7):745-747. doi: 10.1001/jamacardio.2020.1282. No abstract available. PMID 32242890
- [Background] Vaduganathan M, Vardeny O, Michel T, McMurray JJV, Pfeffer MA, Solomon SD. Renin-Angiotensin-Aldosterone System Inhibitors in Patients with Covid-19. N Engl J Med. 2020 Apr 23;382(17):1653-1659. doi: 10.1056/NEJMsr2005760. Epub 2020 Mar 30. No abstract available. PMID 32227760